CLINICAL TRIAL: NCT04931472
Title: Feasibility and Acceptability of the Clinical Frailty Scale in a Swedish Emergency Department Setting
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Daniel Wilhelms, Principal Investigator, University Hospital, Linkoeping
Other Study IDs: 2021-00875FAA
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Frailty
Keywords: Frailty; Geriatric assessment; Emergency service; Feasibility studies; Geriatric emergency medicine
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the feasibility and acceptability of the Clinical Frailty Scale (CFS).

The scale can potentially be adopted for daily use in the Emergency Department (ED) and have been evaluated with regard to feasibility to a certain extent, but have so far not been evaluated in the Swedish emergency care context.

DETAILED DESCRIPTION:
The CFS is introduced and tested as part of a quality-improvement process regarding elderly people within the three Emergency departments (ED) of Region Östergötland.

CFS is a 9-point scale developed within the Canadian Study of Health and Aging, a pictograph and a clinical description aids to assign scores from very fit to terminally ill. The scale enable clinicians to stratify elderly people's degree of frailty with the help of questions and clinical assessment. However, even excellent tools will not be used if they are too difficult or time consuming. The amount of papers addressing issues regarding feasibility and acceptability of the CFS in a clinical ED-setting is still limited, and for Swedish EDs non-existent.

This study is part of a larger research project, data will be collected in three ways:

A. All eligible patients who visit the ED for a period of six weeks will be enrolled, and subsequently assessed with CFS by one of their responsible health-care professionals (i.e. physician, registered nurse or nurse assistant). The number of screened patients divided by the total number of eligible patients will yield the screening rate. Patient- and organisational related characteristics will be collected from the electronic health record.

B. 100 patients will be assessed when someone from the research team is present to enrol patients and clock the assessments. These work shifts will be selected using the online application Research Randomizer, to randomly include all hours of the day as well as eligible health-care professionals. The research-team member will document the time to complete the assessment using CFS, which will give us the screening time.

C. To assess acceptability, health-care professionals will be sent a questionnaire per email, including two reminders. The questionnaire will consist of Likert scales, multiple-choice questions and open textboxes with the aim to explore facilitators and barriers for screening completion.

Primary aim: To explore the feasibility and acceptability of the CFS in a Swedish Emergency care context.

ELIGIBILITY:
Inclusion Criteria:

* Has been in clinical work at the ED for the period of the current study

Exclusion Criteria:

* Unwilling to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Physicians, registered nurses and assistant nurses working in the ED
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Completion rate | During a period of six weeks
  Proportion of completed Clinical Frailty Scale assessments in relation to the number of eligible patients

SECONDARY OUTCOMES:
Duration of time to make the assessment | The assessment will be made in connection with the patient´s first meeting with the care team, i.e. within 1 hour from the patient´s arrival to the ED
  Measured time from that the health care professionals begins to read the instructions until he/she notes the assigned score.
Patient related characteristics correlated to completion rate | From admission to discharge from the Emergency department, up to 24 hours.
  Age, gender, arrival mode, triage priority and discharge destination compared between the screened and not screened patients
Organisational related characteristics correlated to completion rate | From admission to discharge from the Emergency department, up to 24 hours
  Day and time of arrival compared between the screened and not screened patients
Ease of use | Questionnaire that can be answered within five weeks
  The proportion of distributed answers to alternatives 1 (Not at all easy) to 7 (Very easy) to the question: What is your experience of how it is to decide what CFS score a person has ?
Relevance | Questionnaire that can be answered within five weeks
  The proportion of distributed answers to alternatives 1 (Completely irrelevant) to 7 (Very relevant) to the question: How relevant or irrelevant do you experience that it is to use CFS in the emergency department?
Facilitators to perform assessment | Questionnaire that can be answered within five weeks
  Health care professionals descriptions of what facititates performance of frailty assessments, qualitative analysis of the respondents' written answers in a free text box "
Barriers to perform | Questionnaire that can be answered within five weeks
  The proportion of distributed answers to existing alternatives, and qualitative analysis of the respondents' written answers in the free text box "other reason".

CONTACTS AND LOCATIONS:
Locations (1):
- Akutmottagningen US Östergötland, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewis ET, Dent E, Alkhouri H, Kellett J, Williamson M, Asha S, Holdgate A, Mackenzie J, Winoto L, Fajardo-Pulido D, Ticehurst M, Hillman K, McCarthy S, Elcombe E, Rogers K, Cardona M. Which frailty scale for patients admitted via Emergency Department? A cohort study. Arch Gerontol Geriatr. 2019 Jan-Feb;80:104-114. doi: 10.1016/j.archger.2018.11.002. Epub 2018 Nov 8. PMID 30448693
- [Background] Elliott A, Phelps K, Regen E, Conroy SP. Identifying frailty in the Emergency Department-feasibility study. Age Ageing. 2017 Sep 1;46(5):840-845. doi: 10.1093/ageing/afx089. PMID 28541400
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Derived] Horlin E, Munir Ehrlington S, Toll John R, Henricson J, Wilhelms D. Is the clinical frailty scale feasible to use in an emergency department setting? A mixed methods study. BMC Emerg Med. 2023 Oct 26;23(1):124. doi: 10.1186/s12873-023-00894-8. PMID 37880591
- See also: Research Randomizer is a free resource for researchers and students in need of a quick way to generate random numbers or assign participants to experimental conditions — https://www.randomizer.org/